CLINICAL TRIAL: NCT06805734
Title: Natural History With Focus on Oncological Risk Evaluation in Pediatric Patients With PTEN Pathogenic Variants - Observational Study
Brief Title: Natural History With Focus on Oncological Risk Evaluation in Pediatric Patients With PTEN Pathogenic Variants
Acronym: PTEN_Ped
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Azienda Ospedaliera Sant'Anna (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: PTEN_Ped
Record Dates: First submitted 2024-12-10; First posted 2025-02-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: PTEN Hamartoma Syndrome
Keywords: PTEN; PTHS
MeSH Terms: conditions — Hamartoma Syndrome, Multiple

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study in pediatric patientis carryng PTEN pathogenic variants aimed to define oncological risk in children and provide a deeper insight of the clinical course, establishing an updated follow-up protocol.

DETAILED DESCRIPTION:
PTEN is a tumor suppressor gene that was first linked to cancer predisposition syndromes but, in the following years, its phenotypic spectrum has been in continuous evolution and expansion, and nowadays we know that pathogenic variants n this gene may also be found in children presenting with Autism Spectrum Disorder (ASD), and/or DD and macrocephaly, or also with macrocephaly alone. Thus, the term PTEN Hamartoma Tumor Syndrome (PTHS) is now used when referring to PTEN-related conditions.

Nowadays, there is no recognized standard protocol for pediatric follow-up. The screening in mostly single-Centre-based and generally not performed in infancy, with large variability in protocols and timing.

The penetrance, which was previously believed to follow an age-related pattern, nowadays seems rather to be age-specific, as children mainly present macrocephaly and neuropsychiatric problems (DD/ASD), while adults are diagnosed mostly because of gastrointestinal malignancies, breast cancer, thyroid carcinoma or other tumors. However, it is not always true that adult symptoms never occur in PTHS children and, conversely, pediatric signs may also persist through adulthood.

The present study aims to collect PTEN mutated patients and their relatives diagnosed in Italy and followed in different Centers, offering a large pediatric cohort with a full clinical description and trying to provide a deeper insight of the clinical course and oncological manifestations of PTEN-related syndrome; we would like to establish an updated follow-up protocol in order to address all the possible clinical needs of these children.

ELIGIBILITY:
Inclusion Criteria:

* PTEN pathogenic variants (class 4/5 SNV, gene deletion, intragenic duplication/deletion)
* Pediatric patients (<18 years old) and their affected relatives, male/female, all ethnicities
* The legal representative must agree to follow the screening protocol
* Informed consent signed by the legal representative

Exclusion Criteria:

* Refuse to undergo the exams of the protocol assessment at the diagnosis
* PTEN non-pathogenic variants (VOUS or benign/likely benign vatiants)
* No signed informed consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (<18 years of age at enrollment) with pathogenic variants of PTEN genes (gene sequence variant, intragenic deletion/duplication, whole gene deletion) Carrier parents data would also be collected
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Rate of tumor onset in the pediatric subjects with PTEN pathogenic variants | 5 years
  In the 5 years follow-up the subjects must complete annually the provided follow-up. Most of the exams are performed in order to exclude the onset of PTEN-related tumors, in particular:
  * blood tests: thyroid function, renal function, hepatic function, blood count cell exam: screening for thyroid, kidney, liver and intestinal tumors
  * fecal occult blood (FOB): screening for colorectal cancer and polyps
  * dermatological evaluation (at the diagnosis, further evaluations if clinically needed)
  * thyroid US: screening for thyroid tumors
  * abdominal US: screening for kidney, liver and intestinal tumors
  * clinical follow-up (performed either by a geneticist, a pediatrician or a pediatric neurologist): exams evaluation and global monitoring.
  The oncological risk of the patients would be estimated basing on the number of patients who will develop a tumor, benign or malignant, in the 5-years follow-up.
Rate of tumor onset in the adult relatives of the pediatric subjects also carrying the PTEN pathogenic variant | 5 years
  The oncological risk of tumor onset in the pediatric cohort will be compared with that of relatives carrying pathogenic variants.
  Pediatric patients will undergo annual follow-up for the 5 years of the study. Within the same time frame, adult relatives of the index case carrying the same PTEN variant will also be monitored in order to compare oncological risk in adult and pediatric populations and to evaluate phenotypic differences across different stages of life.

SECONDARY OUTCOMES:
Rate of major malformations | 5 years
  Children will be evaluated in order to exclude the presence of major malformations, including:
  * heart malformations: a heart US would be also performed at diagnosis
  * skin anomalies and global examination: a subcutaneous US will be performed if signs of possible peripheral vascular anomalies are present
  * kidney and liver anomalies: those would be also assessed in the abdominal US already planned yearly
  * limbs anomalies: in particular number of fingers/toes and limbs asymmetry
Rate of incidence of brain MRI anomalies | 5 years
  All children will undergo a brain MRI to evaluate the presence or absence of cerebral anomalies
Rate of incidence of neurological comorbidities | 5 years
  The presence or absence of possible neurological comorbidities will be investigated at diagnosis and at every clinical follow-up and data will be recorded in order to estimate the prevalence of the problem in the PTEN cohort.
  Specifically, data about the following issues will be collected:
  * epilepsy
  * clinical neurological signs
  * sleep disorder
  * other neurological comorbidities.
Rate of incidence of neurodevelopmental disorders | 5 years
  The presence or absence of neurodevelopmental diagnosis will be investigated at diagnosis, if not already assessed, and at every clinical follow-up and data will be recorded in order to estimate the prevalence of the problem in the PTEN cohort.
  Global development and/or Intelligence Quotient level will be evaluated with standardized assessment tools, optimized for age and development. Griffiths Mental Development Scale - GMDS, Wechsler Preschool and Primary Scale of Intelligence - WPPSI, Wechsler Intelligence Scale for Children - WISC, and Leiter scales.
  The presence of signs and symptoms of Autism Spectrum Disorder and other possible behavioral problems would also be assessed with standardized tools, both scales (Autism Diagnostic Observation Schedule - ADOS) and questionnaires (Child Behavior Checklist - CBCL, Social Responsiveness Scale - SRS, Adaptive Behavior Assessment System - ABAS).
To analyze Head Circumferences and development of growth HC curves in PTEN patients (data of affected parents will be also recorded) | 5 years
  The HC measures will be monitored at diagnosis at at every follow-up visit in order to follow the head growth of the patients; data about the affected parents will also be recorded. To record data, WHO growth charts will be used as standardized charts.
  Data will be used to develop a PTEN-specific head circumference growth chart.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The participant centers in Italy will share data with the PI Institution. Study protocols and consent forms will be shared with the Institutions collaborating in the study in order to have omogeneous data record.
  Clinicians from the collaborative Centers will return anonymized data to the PI Institution.
Supporting Information: Study Protocol, ICF
Time Frame: 10 years, from August 1st 2024 to July 31st 2034
Access Criteria: Data would be collected and recorded in encrypted Excel sheets with no name/surname/tax code shown; we ensure at each site the accuracy, completeness and timeliness of the files.
  Only the clinical personnel (medical doctors and neuropsychologists) involved in the study will have access to data, that could be accessed anytime but only from the Institutional Organizations participating in the study.
  Data will be stored at Carlo Besta Institute (SSD Sindromi Genetiche con Disabilità Intellettiva e Disturbi dello Spettro Autistico) for 10 years.

REFERENCES:
- [Background] Compton-Smith RN, Fawcett JW. Systemic lupus erythematosus associated with procainamide. Br J Clin Pract. 1967 May;21(5):248-51. No abstract available. PMID 6046409
- [Background] Chen CY, Chen J, He L, Stiles BL. PTEN: Tumor Suppressor and Metabolic Regulator. Front Endocrinol (Lausanne). 2018 Jul 9;9:338. doi: 10.3389/fendo.2018.00338. eCollection 2018. PMID 30038596
- [Background] Rademacher S, Eickholt BJ. PTEN in Autism and Neurodevelopmental Disorders. Cold Spring Harb Perspect Med. 2019 Nov 1;9(11):a036780. doi: 10.1101/cshperspect.a036780. PMID 31427284